CLINICAL TRIAL: NCT01155687
Title: Psychosocial Counseling in Afghanistan
Status: Completed | Type: Observational
Sponsor: University of Konstanz (Other)
Collaborators: European Union (Other)
Responsible Party: Prof. Dr. Thomas Elbert, Sarah Ayoughi, University of Konstanz
Other Study IDs: EuropeAid/127054/C/SER/MULTI
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-06

CONDITIONS: Mental Health; Stress
Keywords: afghanistan; depression; anxiety; social stress; counseling; medication; psychotherapy; mental health
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Psychosocial counseling: the group received annualized treatment of psychosocial counseling
- Medication: this group received medical treatment by the local medical doctor

SUMMARY:
The assessment intends to investigate the efficacy of psychosocial counseling for the treatment of help seeking individuals with psychosocial problems in Mazar-e-Sharif, Afghanistan. Treatment was administered by local counselors who had received specific education and training

DETAILED DESCRIPTION:
Psychosocial stress due to conflict and war causes major mental health problems in many resource-poor countries, especially those coping with ongoing war-like conditions. There is a lack of intervention research in these population. The purpose of this assessment was to examine whether the type of psychosocial counseling developed by our group is effective in reducing symptoms of depression and anxiety and significantly increasing the quality of life of help-seeking Afghans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mental health problems by a local medical doctor

Exclusion Criteria:

* Schizophrenia
* Mental retardation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Afghan people at primary care clinic seeking help because of mental health problems
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HSCL 25 | Symptoms were assessed at baseline
  Symptoms of Depression and Anxiety measured with the HSCL 25
HSCL 25 | 3-month follow-up
  Symptoms of Depression and Anxiety measured with the HSCL 25
HSCL 25 | Assessment at 12-month-follow-up
  Symptoms of Depression and Anxiety measured with the HSCL 25

SECONDARY OUTCOMES:
M.I.N.I. (Mini-International Neuropsychiatric Interview) | Symptoms were assessed at baseline
  To assess, if the patients have a current Major Depression, the depression section from the "Mini-International Neuropsychiatric Interview" (Sheehan, & Janavs, 1998) was included
Psychosocial stressors and coping mechanism | Symptoms were assessed at baseline
  Psychosocial stressors and coping mechanism of the participants were investigated in expert interviews
Screening for Depression | Symptoms were assessed at baseline
  A culturally grounded assessment measure developed in close collaboration with a team of Afghan experts explored current depressive symptoms
M.I.N.I. (Mini-International Neuropsychiatric Interview) | Assessment at 3-month-follow-up
  To assess, if the patients have a current Major Depression, the depression section from the "Mini-International Neuropsychiatric Interview" (Sheehan, & Janavs, 1998) was included
M.I.N.I (Mini-International Neuropsychiatric Interview) | Assessment at 12-month-follow-up
  To assess, if the patients have a current Major Depression, the depression section from the "Mini-International Neuropsychiatric Interview" (Sheehan, & Janavs, 1998) was included
Psychosocial stressors and coping mechanism | Assessment at 3-month-follow-up
  Psychosocial stressors and coping mechanism of the participants were investigated in expert interviews
Psychosocial stressors and coping mechanism | Assessment at 12-month-follow-up
  Psychosocial stressors and coping mechanism of the participants were investigated in expert interviews
Screening for Depression | Assessment at 3-month-follow-up
  A culturally grounded assessment measure developed in close collaboration with a team of Afghan experts explored current depressive symptoms
Screening for Depression | Assessment at 12-month-follow-up
  A culturally grounded assessment measure developed in close collaboration with a team of Afghan experts explored current depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Dr., Principal Investigator — University of Konstanz; Sarah Ayoughi, Principal Investigator — University of Konstanz
Locations (1):
- Counseling Center Mazar-e-Sharif, Mazari Sharif, Balkh, Afghanistan

REFERENCES:
- [Derived] Ayoughi S, Missmahl I, Weierstall R, Elbert T. Provision of mental health services in resource-poor settings: a randomised trial comparing counselling with routine medical treatment in North Afghanistan (Mazar-e-Sharif). BMC Psychiatry. 2012 Feb 29;12:14. doi: 10.1186/1471-244X-12-14. PMID 22375947